CLINICAL TRIAL: NCT01583673
Title: Assessment of Growth of Infants Fed an Amino Acid Based Formula
Brief Title: Growth of Infants Fed an Amino Acid Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 09.56.PED
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2014-06

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amino Acid Formula (Experimental): Hypoallergenic baby formula
  Interventions: Other: Amino Acid Formula
- Amino Acid commercial formula (Active Comparator): Hypoallergenic commercial amino acid formula
  Interventions: Other: Amino Acid formula

INTERVENTIONS:
Other: Amino Acid Formula — Subjects will be fed the assigned study formula from enrollment to 4 months (112 days) of age.Infants will be fed orally, ad libitum with the assigned formula
  Arms: Amino Acid Formula
Other: Amino Acid formula — Subjects will be fed the assigned study formula from enrollment to 4 months (112 days) of age.Infants will be fed orally, ad libitum with the assigned formula
  Arms: Amino Acid commercial formula

SUMMARY:
The primary objective of the clinical trial is to compare growth in infants (expressed as weight gain in g/day) consuming a new Amino Acid Formula to infants consuming a commercially available hypoallergenic formula over a period of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full-term (>= 37 weeks gestation)
* Birth weight between >= 2500 and < =4500 g
* 0-17 days of age on enrolment (day 0 is day of birth)
* Infant's mother has elected not to breastfeed and to exclusively formula-feed infant
* Study explained and written information provided with Caregiver demonstrating understanding of the given information
* Informed consent signed (parent/legal representative)

Exclusion Criteria:

* Congenital illness or malformation that may affect infant feeding and/or normal growth
* Suspected or known allergy to cow's milk protein
* Significant pre-natal and/or post-natal disease
* Any readmission to hospital (except for hyperbilirubinemia) prior to enrolment
* Infant receiving prescription medication (with exception of topical antibiotics and/or treatment for thrush) or frequent use of over the counter medications except vitamin and mineral supplements
* Infant currently participating in another conflicting clinical study
* Infant's family who in the Investigator's assessment cannot be expected to comply with the protocol

Max Age: 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Weight Gain | 4 months
  Mean weight gain (g/day) from enrollment to 4 months of age

SECONDARY OUTCOMES:
tolerance | 4 months
  Tolerance will be evaluated based on formula intake, stool characteristics, vomiting/spitting up and behavior from enrollment to 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Corkins, MD, Principal Investigator — Le Bonheur Children's Hospital
Locations (17):
- United States (17):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Alabama Clinical Therapeutics/Southlake Pediatrics, Birmingham, Alabama
  - Clinical Research Consortium Arizona, Phoenix, Arizona
  - Lutheran General Children's Hospital, Park Ridge, Illinois
  - Nassim, MCMonigle, Mescia and Associates, New Albany, Indiana
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Southwestern Medical Clinic, Niles, Michigan
  - Southwestern Medical Clinic, Stevensville, Michigan
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Blue Ridge Pediatric and Adolescent Medicine, Inc., Boone, North Carolina
  - Haywood Pediatric and Adolescent Medicine Group, P.A., Clyde, North Carolina
  - Tarheel Clinical Research, Raleigh, North Carolina
  - Ohio Pediatric Research Assn., Dayton, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Jean Brown Research, Salt Lake City, Utah
  - Clinical Research Specialists of Utah, Inc, Spanish Fork, Utah

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765